CLINICAL TRIAL: NCT06835738
Title: Implementation of Multiple Micronutrient Supplementation (MMS) for Pregnant Women in Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Vitamin Angels (Unknown); UNICEF (Other); Child and Family Foundation of Uganda (Unknown); Kirk Humanitarian (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00022536/MOD5681
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Nutrient Deficiency

STUDY DESIGN:
Intervention Model Description: MMS will be implemented across 8 districts in Uganda within 3 regions of Uganda. Two regions have 3 study districts/arms and one region (Karamoja) has two study districts/arms. Study arms/districts have been purposively selected.
  * Study Arm 1 (3 districts): Provision of 6 bottles each containing 30 tablets of MMS dispensed monthly over the course of a woman's pregnancy). along with the novel "job aid/adherence calendar"
  * Study Arm 2 (3 districts): Provision of 1 bottle containing 180 tablets dispensed to the pregnant woman attending the first ANC visit; along with the novel "job aid/adherence calendar"
  * Study Arm 3 (2 districts): Provision of 2 bottles each containing 90 tablets of MMS dispensed at two different time points during pregnancy along with the novel "job aid/adherence calendar"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced MMS delivery with six 30-count bottles (standard packaging amount for IFA) (Active Comparator): Pregnant women are provided with six 30-count bottles of MMS monthly during pregnancy, along with the novel job aid/adherence calendar and associated enhanced MMS counseling (1 district within each of the 3 study regions).
  Interventions: Dietary Supplement: Multiple Micronutrient Supplement (MMS) - dispensed in six 30-count bottles
- Enhanced MMS delivery with one 180-count bottle (Active Comparator): Pregnant women are provided with one 180-count bottle of MMS at the first ANC visit, along with the novel job aid/adherence calendar and associated enhanced MMS counseling (1 district within each of the 3 study regions).
  Interventions: Dietary Supplement: Multiple Micronutrient Supplement (MMS) - dispensed in one 180-count bottle
- Enhanced MMS delivery with two 90-count bottles (Active Comparator): Pregnant women are provided with two 90-count bottles of MMS at two different time points during pregnancy, along with the novel job aid/adherence calendar and associated enhanced MMS counseling (1 district within 2 of the study regions (e.g., 2 districts).
  Interventions: Dietary Supplement: Multiple Micronutrient Supplement (MMS) - dispensed in two 90-count bottles

INTERVENTIONS:
Dietary Supplement: Multiple Micronutrient Supplement (MMS) - dispensed in six 30-count bottles — MMS is a daily supplement provided to pregnant women. It will be delivered to pregnant women through the specified bottle-count protocol as designated by the 3 study arms. ANC providers will be trained to counsel pregnant women on using MMS using a novel job aid/adherence calendar.
  Arms: Enhanced MMS delivery with six 30-count bottles (standard packaging amount for IFA)
Dietary Supplement: Multiple Micronutrient Supplement (MMS) - dispensed in one 180-count bottle — MMS is a daily supplement provided to pregnant women. It will be delivered to pregnant women through the specified bottle-count protocol as designated by the 3 study arms. ANC providers will be trained to counsel pregnant women on using MMS using a novel job aid/adherence calendar.
  Arms: Enhanced MMS delivery with one 180-count bottle
Dietary Supplement: Multiple Micronutrient Supplement (MMS) - dispensed in two 90-count bottles — MMS is a daily supplement provided to pregnant women. It will be delivered to pregnant women through the specified bottle-count protocol as designated by the 3 study arms. ANC providers will be trained to counsel pregnant women on using MMS using a novel job aid/adherence calendar.
  Arms: Enhanced MMS delivery with two 90-count bottles

SUMMARY:
The objective of this research is to understand how antenatal multiple micronutrient supplements (MMS) can be effectively implemented and scaled within the Uganda national health system context to support improved maternal nutrition and birth outcomes. Formative research has been conducted to design the implementation strategies that will be tested in this second phase of the study. The objectives are to:

* Describe the implementation of the MMS intervention (which consists of MMS product, a social behavior change communication (SBCC) strategy, capacity building, MMS supply chain support, monitoring, and evaluation) and explore acceptability, feasibility, fidelity, coverage, and potential for sustainability.
* Determine the effect of dispensing MMS in different bottle counts on MMS adherence and ANC attendance among pregnant women.
* Determine the cost and budget impact of MMS intervention implementation integrated in the Ugandan ANC service delivery system

DETAILED DESCRIPTION:
Within the context of the existing antenatal care system, investigators will utilize qualitative and quantitative methods to answer the following research questions:

1. What is the acceptability, feasibility, fidelity, coverage, and potential for sustainability of an MMS intervention that includes MMS product, a contextualized social behavior change communication (SBCC) plan, capacity strengthening, and modified recording and reporting).
2. Does the number of MMS pills in a bottle affect/influence adherence to MMS and/or attendance at ANC attend (30 count bottle vs 90 count bottle vs 180-count bottle).
3. What is the cost and budget impact of implementing MMS intervention within the antenatal care (ANC( service delivery system in Uganda.

This is a 3-arm quasi-experimental implementation research (IR) study utilizing a mixed methods data collection approach across multiple study populations (e.g., national, regional, and district-level decision makers, healthcare providers, pregnant women, and other community members). The three study arms are: Study Arm #1 (MMS 180-count), Study Arm #2 (MMS 30-count) and Study Arm #3 (MMS 90-count).

The IR will be conducted in 8 districts representing the South Central, Acholi, and Karamoja regions of Uganda. Sufficient MMS will be provided to the 8 districts to ensure full implementation of MMS across all government (public) facilities and private not-for-profit (PNFP) facilities within the 8 study districts. In other words, all pregnant women who attend ANC through either a public or PNFP health facility within the 8 study districts will be offered MMS rather than IFA.

Each district will be assigned to receive a specific "bottle-count" to be provided to all pregnant women attending ANC in that district. All women will be provided with 180 tablets of MMS delivered in the "bottle-count" option assigned to the district where she is seeking services. The 3 "bottle-count" options are: 1) 1 bottle containing 180 tablets dispensed to the pregnant woman attending the first ANC visit; 2) 2 bottles each containing 90 tablets of MMS dispensed at two different time points during pregnancy; or 3) 6 bottles each containing 30 tablets of MMS dispensed monthly over the course of a woman's pregnancy). All pregnant women who are assigned to a 30 or 90 bottle count will continue with that bottle count throughout the women's life of pregnancy and postpartum period.

Each "bottle-count" equates to a study arm. Each of the 3 study regions will have slightly different study arms. The districts/study arms within each region were purposively selected under the formative (phase I) of the study. Because there are 3 districts in both the South-Central Region and the Acholi region, each of the 3 districts will serve as a study arm representing one of the three "bottle-count" options. Because there are only 2 districts in the Karamoja region, there will not be a 90-count study-arm.

The study will undertake data collection at approximately 6 facilities per district, representative of the total number of facilities in the districts. Facilities will be purposively selected after being stratified based on the level of the health facility (health center II, health center III, health center IV, or hospital), ownership (government or PNFP), and geographic location.

ELIGIBILITY:
Inclusion Criteria for Pregnant women- Enrolled for follow-up throughout pregnancy (sample 1)

* ≤24 weeks of amenorrhea/gestation as verified by health professionals
* Attending first ANC visit at government or PNFP health facilities.
* Accepted to take MMS at first ANC visit

Exclusion Criteria for Pregnant women- Enrolled for follow-up throughout pregnancy (sample 1)

* Pregnant women with pre-existing hematological conditions such as sickle cell anemia, thalassemia, hemochromatosis.
* Pregnant women planning to relocate outside the study district during the study period.

Inclusion Criteria for Pregnant women / Women that have recently delivered (single contact) (sample 2)

* Currently pregnant woman or a woman who is not more than 8 weeks postpartum.
* Received MMS at an ANC visit at least 3 months ago or more.
* Attended at least any 2 monthly ANC visits.
* Attending/attended ANC at government or private-not-for-profit health facility.

Exclusion Criteria for Pregnant women / Women that have recently delivered (single contact) (sample 2)

* Enrolled in study population 1.
* Women who are more than 8 weeks postpartum.

Inclusion Criteria for ANC providers having ANC health education/counseling with pregnant woman(en) observed (sample 3)

• Healthcare providers that are currently providing ANC health education (group) or ANC individual counseling at government or PNFP health facilities.

Exclusion Criteria for ANC providers having ANC health education/counseling with pregnant woman(en) observed (sample 3) • Healthcare providers that are currently providing ANC health education (group) or ANC individual counseling to a woman(en) that have not provided written informed consent to have the ANC session observed.

Inclusion Criteria for Influential family members (male partners & mothers/mothers-in law) (sample 4)

* Spouse or partner of a pregnant woman or woman with a child less than 8 weeks old who is receiving/ has received ANC services in one of the 8 study districts.
* Mother or mother-in-law of a pregnant woman or woman with a child less than 8 weeks old who is receiving/ has received ANC services in one of the 8 study districts.

Exclusion Criteria for Influential family members (male partners & mothers/mothers-in law) (sample 4) • None

Inclusion Criteria for Healthcare Providers- including facility in-charge, ANC providers, Health Assistants, staff in-charge of records, and stores manager (sample 5)

* Health workers who provide ANC services (e.g., midwives/nurse, medical/ clinical officers, health assistants, and nutrition focal person) at government or private-not-for-profit facilities in one of the 8 study districts.
* Health facility staff (e.g., Facility In-charge, Maternity In-charge, Pharmacy/Stores In-charge) at government or private-not-for-profit facilities in one of the 8 study districts.

Exclusion Criteria for Healthcare Providers- including facility in-charge, ANC providers, Health Assistants, staff in-charge of records, and stores manager (sample 5)

• None

Inclusion Criteria for Community Health Workers (VHTs) and Mentor Mothers (sample 6) • Voluntary Health Team (VHT), Mentor Mothers, or Para-socials attached to at least one of the study facilities.

Exclusion Criteria for Community Health Workers (VHTs) and Mentor Mothers (sample 6) • None

Inclusion Criteria for National, regional, and district-level stakeholders (sample 7)

* National, regional, or district-level decision-makers working in nutrition, maternal, newborn and child health, district health educator or pharmaceutical roles associated with the antenatal care system in Uganda.
* Implementing partners involved in direct implementation of MMS within the 8 study districts

Exclusion Criteria for National, regional, and district-level stakeholders (sample 7)

• None

Inclusion Criteria for Pregnant women - interviewed during post-intervention Household Coverage Survey (sample 8)

* Woman who has been pregnant or delivered within the study period.
* Household is within one of the 4 selected districts.

Exclusion Criteria for Pregnant women - interviewed during post-intervention Household Coverage Survey (sample 8)

• Women who moved to the district after delivery.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4077 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MMS Adherence (amount) as assessed by number of MMS tablets consumed | 3-month post-enrolment, 6-month post-enrolment visit, 6-week postpartum visit
  The number of MMS tablets (from a total possible 180 tablets) a pregnant woman consumes (sample 1).
MMS Adherence (frequency) as assessed by the frequency of tablets consumed | 3-month post-enrolment, 6-month post-enrolment visit, 6-week postpartum visit
  The frequency of which MMS tablets are consumed by a pregnant woman. (sample group 1)
ANC Adherence as assessed by the number of ANC visits throughout pregnancy | 3-month post-enrolment, 6-month post-enrolment visit, 6-week postpartum visit
  The number of ANC visits (from a total possible of 8 visits) a pregnant woman makes throughout her pregnancy (sample 1)

SECONDARY OUTCOMES:
Proportion of pregnant women who indicate MMS Acceptability | 3-month post-enrolment visit, 6-month post-enrolment visit, 6-week postpartum visit
  The proportion of pregnant women (sample group 1 and 2) who agree with domain-specific statements which reflect different aspects of MMS acceptability (MMS packaging, MMS physical properties, MMS side effects, and MMS counseling using The Theoretical Framework of Acceptability uses a 5-point Likert scale where 5 is "strongly agree" and 1 is "strongly disagree". Score range 5-35, a higher score reflects higher acceptability.
MMS Acceptability among Health Providers assessed by focus group discussions | 6 months, 12 months
  Healthcare provider acceptability of MMS across multiple domains (e.g., feasibility of delivering counseling and packaging, time burden) (sample group 5). Measured via focus group discussions at two time points during the study (middle and end).
Fidelity of providing MMS among Health Providers as assessed by focus group discussions | 3-months, 6-months, 9-months, and 12-months
  Administration of an observation checklist (sample group 3) and a Healthcare Provider Survey (sample 5) at 4 time points during the study

OTHER OUTCOMES:
Number of pregnant women being given 180 tablets of MMS | 14 months
  MMS coverage as assessed by the number of pregnant women or recently pregnant women (sample 8) reporting having been given 180 tablets of MMS as compared to the estimated number of pregnant women in the population (e.g., within the 8 study districts) via post-implementation household survey.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Fox, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Lyantonde GH, Lyantonde, Uganda

IPD SHARING:
Plan to Share IPD: No